CLINICAL TRIAL: NCT01616355
Title: Denture Condition: Influence on Masticatory Performance, Volatile Sulfur Compounds and Presence of Biofilm
Brief Title: Evaluation of Sodium Hypochlorite as a Denture Cleanser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Sheila Rodrigues de Sousa Porta, PhD Student, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 068/2008
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Problems With Dentures
Keywords: denture, complete;; sodium hypochlorite;; disinfection;; surface roughness;; color stability.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Sodium hypochlorite immersion — Dentures daily immersion in a 0.5% sodium hypochlorite solution for 3 minutes.

SUMMARY:
The present study tried to integrate all aspects of denture care: patient satisfaction with the treatment, denture decontamination and base material defects after decontamination processing.

DETAILED DESCRIPTION:
Considering that it is necessary to stipulate a simple and effective routine protocol for denture cleaning the aim of this study was to evaluate, in vivo, the efficacy of 0.5% sodium hypochlorite (NaOCl) as a denture cleanser and its effect on color stability and surface roughness of complete dentures. The patients' satisfaction with the denture cleaning method was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* complete denture wearers; adequate general health conditions
* ability to comply with the experimental protocol
* time of denture use: at least one year prior the study
* denture base material: heat-polymerized acrylic resin.

Exclusion Criteria:

* the use of antifungal agents or antiseptic mouthwashes during the pre-experimental and experimental period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Microorganisms reduction | Baseline, 30, 60 and 90 days
  Quantitative analysis of total microorganisms and Candida spp. Samples for culture were collected from dentures and saliva.
Changes in base acrylic resin | Baseline, 30, 60 and 90 days
  Color stability and surface roughness evaluation

SECONDARY OUTCOMES:
Patients' satisfaction with the denture cleaning protocol | 30, 60 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Altair A Del Bel Cury, PhD, Study Chair — School of Dentistry of Piracicaba, State University of Campinas; Sheila RS Porta, PhD Student, Principal Investigator — School of Dentistry of Piracicaba, State University of Campinas
Locations (1):
- School of Dentistry of Piracicaba, UNICAMP, Piracicaba, São Paulo, Brazil